CLINICAL TRIAL: NCT07240103
Title: Blood-Interstitial Fluid Glucose Gap: A Novel Indicator for Assessing Metabolic Status and Mortality Risk in Critically Ill Patients
Brief Title: Blood-Interstitial Fluid Glucose Gap
Status: Completed | Type: Observational
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Other Study IDs: Glucose Gap
Record Dates: First submitted 2025-11-13; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Critical Illness; Metabolism Disorders
Keywords: Glucose Gap; Metabolic Monitoring; Critically Ill Patients; Prognosis; Insulin Resistance
MeSH Terms: conditions — Critical Illness; Metabolic Diseases; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metabolic monitoring is fundamental to guiding nutritional therapy in critically ill patients. Although indirect calorimetry is the established gold standard for measuring resting energy expenditure, its routine clinical use is constrained by practical challenges, including procedural complexity, time-intensive nature, significant cost, and limited feasibility in patients on advanced life support, such as extracorporeal membrane oxygenation (ECMO). Dysregulation of glucose metabolism is common in this population, characterized not only by absolute dysglycemia but also-and perhaps more critically-by impairments in the efficiency of glucose transport and utilization across the microcirculatory continuum (from arterial blood, through the interstitial space, to venous return). This study seeks to examine the relationship between novel dynamic metrics-such as the arterio-interstitial glucose gradient-and key clinical parameters, including energy expenditure, organ function, and patient outcomes. Our objective is to assess the utility of these measures as minimally invasive, real-time biomarkers of metabolic state in critical illness.

DETAILED DESCRIPTION:
This prospective observational study aims to investigate the association between blood-interstitial fluid glucose concentration differences and resting energy expenditure, organ function, and clinical outcomes in critically ill patients, while also exploring potential factors influencing these glucose concentration differences.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years and < 80 years
* ICU stay ≤48 hours
* Expected ICU stay > 24 hours
* APACHE II score≥ 8

Exclusion Criteria:

* local infection within the sensor placement area
* Laparotomy within lower abdomen
* Participated in this study before
* In other clinical trails

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill patient
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
ICU Mortality | From date of study enrollment until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 60 days
  The incidence of all-cause death during the patient's stay in the Intensive Care Unit

SECONDARY OUTCOMES:
Duration of Vasopressor Dependency | From date of study enrollment until the date of vasopressor cessation for at least 24 hours, assessed up to 30 days
  The total length of time a patient requires continuous intravenous vasoactive drugs to maintain adequate blood pressure.
Duration of Invasive Mechanical Ventilation | From date of study enrollment until the date of successful extubation, tracheostomy, or death from any cause, whichever came first, assessed up to 30 days
  The total length of time a patient requires endotracheal intubation and support from a mechanical ventilator.
Duration of Continuous Renal Replacement Therapy (CRRT) | From date of study enrollment until the date of CRRT discontinuation for at least 24 hours or death from any cause, whichever came first, assessed up to 30 days
  The total length of time a patient requires continuous renal replacement therapy for acute kidney injury.

CONTACTS AND LOCATIONS:
Overall Officials: Wenkui Yu, Professor, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Result] Houben AJHM, Martens RJH, Stehouwer CDA. Assessing Microvascular Function in Humans from a Chronic Disease Perspective. J Am Soc Nephrol. 2017 Dec;28(12):3461-3472. doi: 10.1681/ASN.2017020157. Epub 2017 Sep 13. PMID 28904002
- [Result] Gouvea Bogossian E, Taleb C, Aspide R, Badenes R, Battaglini D, Bilotta F, Blandino Ortiz A, Caricato A, Castioni CA, Citerio G, Ferraro G, Martino C, Melchionda I, Montanaro F, Monleon Lopez B, Nato CG, Piagnerelli M, Picetti E, Robba C, Simonet O, Thooft A, Taccone FS. Cerebro-spinal fluid glucose and lactate concentrations changes in response to therapies in patIents with primary brain injury: the START-TRIP study. Crit Care. 2023 Mar 31;27(1):130. doi: 10.1186/s13054-023-04409-6. PMID 37004053
- [Result] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Hylander Moller M, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock 2021. Crit Care Med. 2021 Nov 1;49(11):e1063-e1143. doi: 10.1097/CCM.0000000000005337. No abstract available. PMID 34605781
- [Result] Nuyttens L, Heyerick M, Heremans G, Moens E, Roes M, Van Dender C, De Bus L, Decruyenaere J, Dewaele J, Vandewalle J, Libert C. Unraveling mitochondrial pyruvate dysfunction to mitigate hyperlactatemia and lethality in sepsis. Cell Rep. 2025 Aug 26;44(8):116032. doi: 10.1016/j.celrep.2025.116032. Epub 2025 Jul 21. PMID 40694477
- [Result] Jaiswal N, Gavin MG, Quinn WJ 3rd, Luongo TS, Gelfer RG, Baur JA, Titchenell PM. The role of skeletal muscle Akt in the regulation of muscle mass and glucose homeostasis. Mol Metab. 2019 Oct;28:1-13. doi: 10.1016/j.molmet.2019.08.001. Epub 2019 Aug 5. PMID 31444134
- [Result] Marik PE, Bellomo R. Stress hyperglycemia: an essential survival response! Crit Care Med. 2013 Jun;41(6):e93-4. doi: 10.1097/CCM.0b013e318283d124. No abstract available. PMID 23685597
- [Result] Mahdavi S, Anthony NM, Sikaneta T, Tam PY. Perspective: Multiomics and Artificial Intelligence for Personalized Nutritional Management of Diabetes in Patients Undergoing Peritoneal Dialysis. Adv Nutr. 2025 Mar;16(3):100378. doi: 10.1016/j.advnut.2025.100378. Epub 2025 Jan 20. PMID 39842720
- [Result] Achamrah N, Delsoglio M, De Waele E, Berger MM, Pichard C. Indirect calorimetry: The 6 main issues. Clin Nutr. 2021 Jan;40(1):4-14. doi: 10.1016/j.clnu.2020.06.024. Epub 2020 Jul 2. PMID 32709554
- [Result] De Waele E, van Zanten ARH. Routine use of indirect calorimetry in critically ill patients: pros and cons. Crit Care. 2022 May 5;26(1):123. doi: 10.1186/s13054-022-04000-5. No abstract available. PMID 35513872
- [Result] Moonen HPFX, Beckers KJH, van Zanten ARH. Energy expenditure and indirect calorimetry in critical illness and convalescence: current evidence and practical considerations. J Intensive Care. 2021 Jan 12;9(1):8. doi: 10.1186/s40560-021-00524-0. PMID 33436084
- [Result] Graf S, Karsegard VL, Viatte V, Heidegger CP, Fleury Y, Pichard C, Genton L. Evaluation of three indirect calorimetry devices in mechanically ventilated patients: which device compares best with the Deltatrac II((R))? A prospective observational study. Clin Nutr. 2015 Feb;34(1):60-5. doi: 10.1016/j.clnu.2014.01.008. Epub 2014 Jan 21. PMID 24485773
- [Result] Lakenman PLM, van der Hoven B, van Bommel J, Olieman JF, Joosten KFM. The usefulness of a new indirect calorimeter in critically ill adult patients. Clin Nutr. 2024 Oct;43(10):2267-2272. doi: 10.1016/j.clnu.2024.07.048. Epub 2024 Aug 7. PMID 39208718
- [Result] de Goes CR, Berbel-Bufarah MN, Sanches AC, Xavier PS, Balbi AL, Ponce D. Poor Agreement between Predictive Equations of Energy Expenditure and Measured Energy Expenditure in Critically Ill Acute Kidney Injury Patients. Ann Nutr Metab. 2016;68(4):276-84. doi: 10.1159/000446708. Epub 2016 Jun 10. PMID 27288392
- [Result] Harris JA, Benedict FG. A Biometric Study of Human Basal Metabolism. Proc Natl Acad Sci U S A. 1918 Dec;4(12):370-3. doi: 10.1073/pnas.4.12.370. No abstract available. PMID 16576330
- [Result] Zusman O, Theilla M, Cohen J, Kagan I, Bendavid I, Singer P. Resting energy expenditure, calorie and protein consumption in critically ill patients: a retrospective cohort study. Crit Care. 2016 Nov 10;20(1):367. doi: 10.1186/s13054-016-1538-4. PMID 27832823
- [Result] Singer P, Bendavid I, BenArie I, Stadlander L, Kagan I. Feasibility of achieving different protein targets using a hypocaloric high-protein enteral formula in critically ill patients. Crit Care. 2021 Jun 11;25(1):204. doi: 10.1186/s13054-021-03625-2. PMID 34116714
- [Result] Allingstrup MJ, Kondrup J, Wiis J, Claudius C, Pedersen UG, Hein-Rasmussen R, Bjerregaard MR, Steensen M, Jensen TH, Lange T, Madsen MB, Moller MH, Perner A. Early goal-directed nutrition versus standard of care in adult intensive care patients: the single-centre, randomised, outcome assessor-blinded EAT-ICU trial. Intensive Care Med. 2017 Nov;43(11):1637-1647. doi: 10.1007/s00134-017-4880-3. Epub 2017 Sep 22. PMID 28936712
- [Result] Arabi YM, Casaer MP, Chapman M, Heyland DK, Ichai C, Marik PE, Martindale RG, McClave SA, Preiser JC, Reignier J, Rice TW, Van den Berghe G, van Zanten ARH, Weijs PJM. The intensive care medicine research agenda in nutrition and metabolism. Intensive Care Med. 2017 Sep;43(9):1239-1256. doi: 10.1007/s00134-017-4711-6. Epub 2017 Apr 3. PMID 28374096